CLINICAL TRIAL: NCT04636866
Title: The Prevalence of Helicobacter Pylori Infection in Patients With Peptic Ulcer Disease in Shanghai, 2013 to 2019
Brief Title: The Prevalence of Helicobacter Pylori in Shanghai, 2013 to 2019
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Doctor, Shanghai Jiao Tong University School of Medicine
Other Study IDs: shrj202010171
Record Dates: First submitted 2020-11-14; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Peptic Ulcer; Helicobacter Pylori Infection
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric ulcer
  Interventions: Other: NO intervention
- Duodenal ulcer
  Interventions: Other: NO intervention

INTERVENTIONS:
Other: NO intervention — NO intervention

SUMMARY:
The study was a cross-sectional single-center study, conducted at Renji Hospital, Shanghai Jiaotong university school of medicine. We retrieved the medical records of all patients who had undergone upper gastrointestinal endoscopy from January 1, 2013 through December 31, 2019. The medical records were analyzed for the prevalence of H. pylori infection in patients with peptic ulcers.

ELIGIBILITY:
Inclusion Criteria:

All patients who had undergone upper gastrointestinal endoscopy in Renji Hospital because of uninvestigated dyspepsia during 2013 and 2019 were analyzed.

Exclusion Criteria:

Patients that underwent upper endoscopy for reasons other than uninvestigated dyspepsia such as cirrhosis follow-up, major systemic diseases or other indications were excluded. Exclusions also included absence of biopsies, unknown H. pylori status and acute ulcer bleeding.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We retrieved the medical records of all patients who had undergone upper gastrointestinal endoscopy because of uninvestigated dyspepsia from January 1, 2013 through December 31, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
the prevalence of Helicobacter pylori and peptic ulcer | 2013.1.1-2019.12.31
  the trends change from 2013 to 2019
the ration of Helicobacter pylori positive peptic ulcers | 2013.1.1-2019.12.31
  the trends change from 2013 to 2019

CONTACTS AND LOCATIONS:
Overall Officials: HONG LU, PhD, Study Director — RenJi Hospital
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No